CLINICAL TRIAL: NCT02852577
Title: Long-term, Open, Naturalistic, Randomized Clinical Trial With Clonazepam and Paroxetine in Panic Disorder With or Without Agoraphobia
Brief Title: Long Term Treatment of Panic Disorder With Clonazepam or Paroxetine
Acronym: LTTPANIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rafael Christophe da Rocha Freire, MD, PhD. Assistant professor., Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0003.0.249.000-09
Record Dates: First submitted 2016-07-21; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: panic disorder; agoraphobia; clonazepam; paroxetine
MeSH Terms: conditions — Panic Disorder; Agoraphobia | interventions — Clonazepam; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonazepam (Active Comparator): Treatment with clonazepam
  Interventions: Drug: Clonazepam
- Paroxetine (Active Comparator): Treatment with paroxetine
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Clonazepam — Administration of clonazepam once a day, flexible dose (0.5 - 2 mg/day), for 36 months. If no remission after 8 weeks augmentation with paroxetine once a day, flexible dose (10 - 40 mg/day), for 34 months.
  Arms: Clonazepam
Drug: Paroxetine — Administration of paroxetine once a day, flexible dose (10 - 40 mg/day), for 36 months. If no remission after 8 weeks augmentation with clonazepam once a day, flexible dose (0.5 - 2 mg/day), for 34 months.
  Arms: Paroxetine

SUMMARY:
The purpose of this study was to determine whether clonazepam and paroxetine are effective in the treatment of panic disorder. Efficacy was evaluated in short-term, long-term and post-treatment.

DETAILED DESCRIPTION:
The current study consisted of three steps. The first step was a naturalistic, prospective, randomized, open clinical trial with clonazepam and paroxetine. Subjects received either flexible dose clonazepam (0.5 - 2 mg/day) or paroxetine (10 - 40 mg/day), in monotherapy for eight weeks. In the second step, those who responded to monotherapy in the short-term study continued with the same drug and dose. Partial responders or non-responders were invited to receive combined pharmacological treatment with clonazepam and paroxetine. Patients received the maximum tolerated doses of clonazepam and paroxetine. The doses were flexible, ranging from 0.5 to 2 mg/day for clonazepam and from 10 to 40 mg/day of paroxetine. All patients were treated for 34 months in the second step. Patients who completed the second step and were in remission were included in the third step. For a period of four months all medications were tapered off. These patients were followed for 6 years with evaluations once a year. Those who relapsed were treated on a naturalistic basis, with drugs or psychotherapy.

This study was conducted in accordance with the ethical principles established by the Declaration of Helsinki and the Brazilian National Ethics Committee (Conselho Nacional de Ética em Pesquisa - CONEP) guidelines. The local Ethics Committee approved the study protocol. Written informed consent was obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of panic disorder, with or without agoraphobia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, text revision (DSM-IV-TR) criteria, as determined by a structured clinical interview.
* At least two panic attacks in the week preceding their inclusion in the study.

Exclusion Criteria:

* Patients unable or unwilling to provide written informed consent.
* Did not complete all the evaluations before study initiation.
* Had comorbidities that could affect clinical evaluation including drug abuse, neurological disorders, or severe personality disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2000-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Severity scores at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Clinical Global Impression Severity scores at 36 months | 36 months
Clinical Global Impression Severity scores at 4 years | 4 years
Clinical Global Impression Severity scores at 9 years | 9 years
Change from baseline of Clinical Global Impression Severity (CGI-S) scale scores at 8 weeks | Baseline, 8 weeks
Change from baseline of Clinical Global Impression Severity (CGI-S) scale scores at 36 months | Baseline, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael C Freire, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Instituto de Psiquiatria da Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nardi AE, Valenca AM, Freire RC, Mochcovitch MD, Amrein R, Sardinha A, Levitan MN, Nascimento I, de-Melo-Neto VL, King AL, de O E Silva AC, Veras AB, Dias GP, Soares-Filho GL, da Costa RT, Mezzasalma MA, de Carvalho MR, de Cerqueira AC, Hallak JE, Crippa JA, Versiani M. Psychopharmacotherapy of panic disorder: 8-week randomized trial with clonazepam and paroxetine. Braz J Med Biol Res. 2011 Apr;44(4):366-73. doi: 10.1590/s0100-879x2011007500020. Epub 2011 Feb 18. PMID 21344132
- [Result] Nardi AE, Valenca AM, Freire RC, Amrein R, Sardinha A, Levitan MN, Nascimento I, de-Melo-Neto VL, King AL, de O e Silva AC, Veras AB, Dias GP, Soares-Filho GL, da Costa RT, Mezzasalma MA, de Carvalho MR, de Cerqueira AC, Hallak JE, Crippa JA, Versiani M. Randomized, open naturalistic, acute treatment of panic disorder with clonazepam or paroxetine. J Clin Psychopharmacol. 2011 Apr;31(2):259-61. doi: 10.1097/JCP.0b013e318210b4ee. No abstract available. PMID 21364347
- [Result] Nardi AE, Freire RC, Mochcovitch MD, Amrein R, Levitan MN, King AL, Valenca AM, Veras AB, Paes F, Sardinha A, Nascimento I, de-Melo-Neto VL, Dias GP, E Silva AC, Soares-Filho GL, da Costa RT, Mezzasalma MA, de Carvalho MR, de Cerqueira AC, Hallak JE, Crippa JA, Versiani M. A randomized, naturalistic, parallel-group study for the long-term treatment of panic disorder with clonazepam or paroxetine. J Clin Psychopharmacol. 2012 Feb;32(1):120-6. doi: 10.1097/JCP.0b013e31823fe4bd. PMID 22198456